CLINICAL TRIAL: NCT03640143
Title: Effectiveness of Various Environmental Measures to Eliminate the Risks of Lead Exposure in Infant Lead Poisoning
Brief Title: Effectiveness of Environmental Measures to Eliminate the Risks of Lead Exposure in Infant Lead Poisoning
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-51
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Poisoning
MeSH Terms: conditions — Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: children with clinical expression of lead poisoning data about venous blood lead will be reported
  Interventions: Other: venous blood lead

INTERVENTIONS:
Other: venous blood lead — data about ve,nous blood lead

SUMMARY:
Infant lead poisoning is the clinical expression of lead poisoning. This environmental disease, still present in France, is the only notifiable non-infectious disease.

Its complications include, in the foreground, disorders of psychomotor development but also include in adults the attack of other systems.

The fight against lead poisoning mainly involves the removal of lead sources. Several methods of eviction exist: a modification of the practices, a palliative rehabilitation, a definitive rehabilitation and a relocation. The effectiveness of each method is not documented. This study therefore aims to compare the effectiveness of these various measures to eliminate the risk of exposure to lead on blood lead.

This study uses the methodology of a multicenter historical cohort. It will begin in the second quarter of 2017. The research centers will be child-environment consultations and mother-child PASS in Avignon, Manosque, Marseille, Nice and Toulon.

The study will be offered to all children monitored in these centers since 2011. The inclusion criteria will include: age <18 years, at least one blood lead ≥ 50μg.L-1, residence declared in PACA and absence opposition. The retrospective data will be incorporated into the prospective monitoring. The necessary number is at least 165 cases of infantile lead poisoning (of which 33 per type of intervention). The primary endpoint will be the kinetics of quarterly venous blood lead. The smallest clinically significant difference in blood lead levels will be 50μg.L-1 between the different groups.

Statistical analysis will use intra- and inter-individual variability analysis by compartmental modeling of the pharmacokinetics of blood lead. An interim analysis will be conducted in 2017 on the retrospective data to confirm the necessary staffing.

DETAILED DESCRIPTION:
Infant lead poisoning is the clinical expression of lead poisoning. This environmental disease, still present in France, is the only notifiable non-infectious disease.

Its complications include, in the foreground, disorders of psychomotor development (behavioral disorders, attention, memory ...) but also include in adults the attack of other systems (kidney disorders, fertility disorders and complications). obstetric).

The fight against lead poisoning mainly involves the removal of lead sources. Several methods of eviction exist: a modification of the practices, a palliative rehabilitation, a definitive rehabilitation and a relocation. The effectiveness of each method is not documented. This study therefore aims to compare the effectiveness of these various measures to eliminate the risk of exposure to lead on blood lead.

Material and methods: This study uses the methodology of a multicenter historical cohort. It will begin in the second quarter of 2017. The research centers will be child-environment consultations and mother-child PASS in Avignon, Manosque, Marseille, Nice and Toulon.

The study will be offered to all children monitored in these centers since 2011. The inclusion criteria will include: age <18 years, at least one blood lead ≥ 50μg.L-1, residence declared in PACA and absence opposition. The retrospective data will be incorporated into the prospective monitoring. The necessary number is at least 165 cases of infantile lead poisoning (of which 33 per type of intervention). The primary endpoint will be the kinetics of quarterly venous blood lead. The smallest clinically significant difference in blood lead levels will be 50μg.L-1 between the different groups.

Statistical analysis will use intra- and inter-individual variability analysis by compartmental modeling of the pharmacokinetics of blood lead. An interim analysis will be conducted in 2017 on the retrospective data to confirm the necessary staffing.

ELIGIBILITY:
Inclusion Criteria:

* minor (under 18 years old),
* AND having at least one blood lead ≥ 50 μg / l between 1/11/2011 and 31/12/2022,
* AND with at least a subsequent check of blood lead,
* AND having been seen at least once by a Child-Environment Consultation or a mother-child PASS in PACA,
* AND declared resident in PACA,

Exclusion Criteria:

* Patient:

  * with no blood lead ≥ 50 μg / l
  * OR adult at the time of diagnosis
  * OR opposed to participation (opposition of a parent or child served by mail)
  * OR without subsequent monitoring of blood lead,
  * OR declared resident outside Paca,
  * OR for which an environmental intervention was carried out at an unknown date
  * OR without a source of exposure found in France (eg first-time migrant child).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: childrem presenting clinical characteristic of poisoning
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
venous blood lead | 3 years
  the kinetics of venous blood lead. The monitoring rhythm is recommended every 3 months in a medical analysis laboratory. The smallest clinically significant difference will be a decrease in blood lead level of 50 μg / l.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publiquye Des Hopitaux de Marseille, Marseille, PACA, France